CLINICAL TRIAL: NCT06923774
Title: A European Multi-Center, Prospective, Single-Arm, Observational Study to Evaluate Real-World Outcomes for the Ion Endoluminal System
Brief Title: European Real-World Registry for Use of the Ion Endoluminal System
Status: Recruiting | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: 1147383C
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Nodule; Lung Cancer
Keywords: Biopsy; Bronchoscopy; pulmonary biopsy; pulmonary nodule localization
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Observation Group: Subjects with biopsy and/or localization of lung nodule(s)
  Interventions: Device: Ion endoluminal system

INTERVENTIONS:
Device: Ion endoluminal system — Lung nodule biopsy and/or localization procedure using the Ion endoluminal system per sites' standard of care

SUMMARY:
The objective of this study is to collect collect real-world data for the Ion endoluminal system.

DETAILED DESCRIPTION:
This is a prospective, observational, multi-center, single-arm study to collect real-world data evaluating procedural characteristics and short- and long-term clinical outcomes following the use of the CE-marked Ion endoluminal system for elective lung nodule biopsies and/or localization procedures. It is a post-market study using the device per the approved indications. All patients will be enrolled per the protocol eligibility criteria. Enrollment for this study will conclude when approximately 1,200 patients have had a nodule biopsy and/or localization procedure attempted or performed.

ELIGIBILITY:
Inclusion Criteria:

* Patient is aged 18 years or older at time of consent.
* Patient is planned to undergo a lung lesion biopsy(s) and/or localization procedure(s) utilizing the Ion endoluminal system.
* Patient is willing and able to give written informed consent for clinical study participation.

Exclusion Criteria:

* Patient is participating in an interventional research study or research study with investigational agents with an unknown safety profile that would interfere with participation in this study or study results.
* Female patient that is pregnant or breast feeding as determined by standard site practices.
* Patient is legally incapacitated or in a legal/court ordered institution or is part of a known vulnerable population, including but not limited to dependency on the sponsor, hospital or study doctor.
* Patient is not willing to comply with post-procedure study participation requirements.
* Investigator, in their professional opinion, has decided that it is in the patient's best interest to not participate in the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planned for an elective lung nodule biopsy and/or localization procedure using the Ion endoluminal system as their standard of care
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Yield | Intra-procedure through 24 month post-procedure
  Diagnostic Yield defined as the sum of true positives and true negatives divided by the total number of nodules biopsied. Primary outcome analyses will exclude subjects that are enrolled for localization procedure only.

SECONDARY OUTCOMES:
Pneumothorax | Intra-procedure through 30 days post-procedure
  Defined as the incidence of subjects that undergo an Ion procedure with a pneumothorax event, requiring intervention
Bleeding | Intra-procedure through the 30 day post-procedure
  Defined as the incidence of subjects that undergo an Ion Procedure with a bleeding event, with a grade of greater than 2 on the Nashville Scale

CONTACTS AND LOCATIONS:
Locations (4):
- Hôpital Marie Lannelongue, Le Plessis-Robinson, France
- Universitätsspital Zürich, Zurich, Switzerland
- United Kingdom (2):
  - University College London Hospitals NHS Foundation Trust, London
  - Wythenshawe Hospital, Manchester University NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No